CLINICAL TRIAL: NCT00145301
Title: A 52-week, International, Multi-center, Randomized, Double-blind, Double-dummy, Parallel-group Clinical Trial to Compare Retention on Treatment, Safety, Tolerability and Efficacy of Lumiracoxib 100 mg od, Lumiracoxib 100 mg Bid and Celecoxib 200 mg od in Patients With Primary Osteoarthritis of Hip, Knee, Hand or Spine
Brief Title: 52 Week, International, Multi-center, Randomized, Double-blind, Double-dummy, Parallel-group Clinical Trial to Compare Retention on Treatment, Safety, Tolerability & Efficacy of Lumiracoxib 100 mg od, Lumiracoxib 100 mg Bid & Celecoxib 200 mg od in Pts With Primary OA of Hip, Knee, Hand or Spine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2369
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, lumiracoxib, retention on treatment, efficacy, safety
MeSH Terms: conditions — Osteoarthritis | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This trial will compare the retention on treatment (based on the rate of patients staying on treatment for 1 year) of patients suffering from primary osteoarthritis using two different doses of lumiracoxib (100 mg od or 100 mg bid) or using celecoxib (200 mg od)

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis in the hip, knee, hand, or spine
* Requiring NSAID therapy

Exclusion Criteria:

* Secondary OA with history and/ or any evidence of the following diseases: rheumatoid arthritis, uncontrolled gout, inflammatory joint disease, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary osteochondromatosis, heritable disorders (e.g. hypermobility), collagen gene mutations, primary fibromyalgia (secondary fibromyalgia is allowed if in the opinion of the investigator it will not interfere with the patient's OA pain assessment), and systemic lupus erythematosus
* History and/ or any evidence of the following diseases in the target joint: septic arthritis, gout, recurrent episodes of pseudogout, Paget's disease of the bone, and articular fracture. If the patient has history of these conditions, then patient should only be excluded if the target joint is affected.
* History of severe adverse reactions of any kind under lumiracoxib or celecoxib treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 3036
Dates: Start 2004-09; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To show that either regimen of lumiracoxib (100mg od or 100mg bid) is not inferior to celecoxib 200mg od with respect to retention rate at 1 year in pts suffering from primary OA in hip, knee, hand or spine.

SECONDARY OUTCOMES:
Safety & tolerability of pts using lumiracoxib vs pts using celecoxib
Efficacy of lumiracoxib vs celecoxib with respect to Patient's assessment of OA pain, Patient's global assessment of disease activity, and Physician's global assessment of disease activity
To compare reasons for discontinuation from treatment with lumiracoxib vs treatment with celecoxib
To validate the psychometric properties of the Short Arthritis assessment Scale (SAS) by analyzing pt reported outcomes collected in this study

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis, Nuremberg, Germany

REFERENCES:
- [Derived] Fleischmann R, Tannenbaum H, Patel NP, Notter M, Sallstig P, Reginster JY. Long-term retention on treatment with lumiracoxib 100 mg once or twice daily compared with celecoxib 200 mg once daily: a randomised controlled trial in patients with osteoarthritis. BMC Musculoskelet Disord. 2008 Mar 7;9:32. doi: 10.1186/1471-2474-9-32. PMID 18328090